CLINICAL TRIAL: NCT00273364
Title: Hematopoietic Stem Cell Therapy for Patients With Inflammatory Multiple Sclerosis Failing Alternate Approved Therapy: A Randomized Study
Brief Title: Stem Cell Therapy for Patients With Multiple Sclerosis Failing Alternate Approved Therapy- A Randomized Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Uppsala University (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DI MS.Randomized2004; NCT03133403 (obsolete NCT alias)
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: stem cell, autoimmune disease, multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hematopoietic Stem Cell Transplantation (Experimental): Hematopoietic Stem Cell Therapy will be performed as follows: Autologous stem cells will be infused after conditioning with Cyclophosphamide and rATG
  Interventions: Procedure: Hematopoietic Stem Cell Therapy
- Standard therapy for MS (Active Comparator): Standard treatment with a conventional drug is the treatment with one of the following drugs: Avonex (interferon beta 1a), Betaseron (interferon beta 1b), Copaxone (glatiramer acetate), Aubagio (teriflunomide), Tysabri (natalizumab), Gilenya (fingolimod) or Dimethyl fumarate (Tecfidera or BG-12)
  Interventions: Drug: Standard treatment with a conventional drug

INTERVENTIONS:
Procedure: Hematopoietic Stem Cell Therapy — After mobilization and harvest of stem cells, stem cells will be infused following conditioning regimen
  Other Names: stem cell infusion
  Arms: Hematopoietic Stem Cell Transplantation
Drug: Standard treatment with a conventional drug — Standard treatment with a conventional drug is the treatment with one of the following drugs: Avonex (interferon beta 1a), Betaseron (interferon beta 1b), Copaxone (glatiramer acetate), Aubagio (teriflunomide), Tysabri (natalizumab), or Gilenya (fingolimod)
  Other Names: standard of care
  Arms: Standard therapy for MS

SUMMARY:
Multiple sclerosis (MS) is at onset an immune-mediated demyelinating disease. In most cases, it starts as a relapsing-remitting disease with distinct attacks and no symptoms between flares. Over years or decades, virtually all cases transition into a progressive disease in which insidious and slow neurologic deterioration occurs with or without acute flares. Relapsing-remitting disease is often responsive to immune suppressive or modulating therapies, while immune based therapies are generally ineffective in patients with a progressive clinical course. This clinical course and response to immune suppression, as well as neuropathology and neuroimaging studies, suggest that disease progression is associated with axonal atrophy. Disability correlates better with measures of axonal atrophy than immune mediated demyelination. Therefore, immune based therapies, in order to be effective, need to be started early in the disease course while MS is predominately an immune-mediated and inflammatory disease. While current immune based therapies delay disability, no intervention has been proven to prevent progressive disability. We propose, as a randomized study, autologous unmanipulated PBSCT using a conditioning regimen of cyclophosphamide and rabbit antithymocyte globulin (rATG) versus FDA approved standard of care (i.e. interferon, glatiramer acetate, mitoxantrone, natalizumab, fingolimod, or tecfidera) in patients with inflammatory (relapsing) MS despite treatment with alternate approved therapy.

DETAILED DESCRIPTION:
To assess the efficacy of autologous PBSCT versus FDA approved standard of care ( i.e. interferon, glatiramer acetate, mitoxantrone, natalizumab, fingolimod, or tecfidera) for inflammatory multiple sclerosis (MS) failing failing alternate approved therapy. The endpoints to be considered in this study are:

2.1 Primary Endpoint:

Disease progression, defined as a 1 point increase in the Expanded Disability Status Scale (EDSS) on consecutive evaluations at least 6 months apart and not due to a non-MS disease process. Patients will be followed for 5 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age between18-55, inclusive.
2. Diagnosis of MS using revised McDonald criteria of clinically definite MS (Appendix I).
3. An EDSS score of 2.0 to 6.0 (Appendix II).
4. Inflammatory disease despite treatment with standard disease modifying therapy including at least 6 months of interferon or copaxone. Inflammatory disease is defined based on both MRI (gadolinium enhancing lesions) and clinical activity (acute relapses *treated with IV or oral high dose corticosteroids and prescribed by a neurologist). Minimum disease activity required for failure is defined as: a) two or more *steroid treated clinical relapses with documented new objective signs on neurological examination documented by a neurologist within the year prior to the study, or b) one *steroid treated clinical relapse within the year prior to study and evidence on MRI of active inflammation (i.e., gadolinium enhancement) within the last 12 months on an occasion separate from the clinical relapse (3 months before or after the clinical relapse).

   * A steroid treated relapse will include a relapse that was severe enough to justify treatment but due to patient intolerance of steroids, or a history of non-response to steroids, they were offered but not used.

Exclusion Criteria**

1. Any illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy.
2. Prior history of malignancy except localized basal cell, squamous skin cancer or carcinoma in situ of the cervix. Other malignancies for which the patient is judged to be cured, such as head and neck cancer, or breast cancer will be considered on an individual basis.
3. Positive pregnancy test
4. Inability or unwillingness to pursue effective means of birth control from the time of evaluation for eligibility until 6 months posttransplant (if on transplant) or until appropriate for non-transplant treatment (if on control arm). Effective birth control is defined as 1) abstinence defined as refraining from all acts of vaginal intercourse; 2) consistent use of birth control pills; 3) injectable birth control methods (Depo-provera, Norplant); 4) tubal sterilization or male partner who has undergone vasectomy; 5) placement of an intrauterine device (IUD); or 6) use, with every act of intercourse, of diaphragm with contraceptive jelly and/or condoms with contraceptive foam.
5. Failure to willingly accept or comprehend irreversible sterility as a side effect of therapy
6. Forced expiratory volume at one second (FEV1) / forced vital capacity (FVC) < 60% of predicted after bronchodilator therapy (if necessary)
7. Diffusing capacity of lung for carbon monoxide (DLCO) < 50% of predicted (for the transplant arm)
8. Resting left ventricular ejection fraction (LVEF) < 50 %
9. Bilirubin > 2.0 mg/dl
10. Serum creatinine > 2.0 mg/dl
11. Known hypersensitivity to mouse, rabbit, or E. Coli derived proteins, or to iron compounds/medications
12. Presence of metallic objects implanted in the body that would preclude the ability of the patient to safely have MRI exams
13. Diagnosis of primary progressive MS
14. Diagnosis of secondary progressive MS
15. Platelet count < 100,000/ul, white blood cell count (WBC) < 1,500 cells/mm3
16. Psychiatric illness, mental deficiency or cognitive dysfunction making compliance with treatment or informed consent impossible
17. Active infection except asymptomatic bacteriuria
18. Use of natalizumab (Tysabri) within the previous 6 months
19. Use of fingolimod (Gilenya) within the previous 3 months
20. Use of teriflunomide (Aubagio) within the previous 2 years unless cleared from the body (plasma concentration < 0.02mcg/ml) following elimination from the body with cholestyramine 8g three times a day for 11 days
21. Prior treatment with CAMPATH (alemtuzumab)
22. Prior treatment with mitoxantrone
23. Any hereditary neurological disease such as Charcot-Marie-Tooth disease (CMT) or Spinocerebellar ataxia (SCA) are contraindications
24. Use of tecfidera within the previous 3 months

    * For patients who clearly have inflammatory disease, an exception can be made if agreed upon by study PI and at least two study neurologists.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2005-11-16 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Result] Burt RK, Balabanov R, Burman J, Sharrack B, Snowden JA, Oliveira MC, Fagius J, Rose J, Nelson F, Barreira AA, Carlson K, Han X, Moraes D, Morgan A, Quigley K, Yaung K, Buckley R, Alldredge C, Clendenan A, Calvario MA, Henry J, Jovanovic B, Helenowski IB. Effect of Nonmyeloablative Hematopoietic Stem Cell Transplantation vs Continued Disease-Modifying Therapy on Disease Progression in Patients With Relapsing-Remitting Multiple Sclerosis: A Randomized Clinical Trial. JAMA. 2019 Jan 15;321(2):165-174. doi: 10.1001/jama.2018.18743. PMID 30644983
- [Derived] Burman J, Fransson M, Totterman TH, Fagius J, Mangsbo SM, Loskog AS. T-cell responses after haematopoietic stem cell transplantation for aggressive relapsing-remitting multiple sclerosis. Immunology. 2013 Oct;140(2):211-9. doi: 10.1111/imm.12129. PMID 23721329

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation | Standard Therapy for MS
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hematopoietic Stem Cell Transplantation | Standard Therapy for MS | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Median (Full Range); unit: years] | 35.6 [18 to 54] | 35.6 [19 to 52] | 35.6 [18 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 39 | 73
  Male | 21 | 16 | 37
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — The EDSS provides a total disability score on a scale that ranges from 0 (no disability) to 10 (worst neurologic disability). Population: The number analyzed in rows differs from the overall enrolled because EDSS were not analyzed on patients who did not receive intervention or who were lost to follow up.
  units on a scale
    number analyzed (Participants) | 52 | 54 | 106
    (all) | 3.4 (1.2) | 3.3 (1.0) | 3.35 (.05)

OUTCOME MEASURES:

1. Primary Outcome: Expanded Disability Status Scale (EDSS) Improvement
Description: The EDSS scale ranges from 0 to 10 in 0.5 increments that represent higher levels of disability. Improvement in EDSS is defined by both a 0.5 or 1.0 points sustained for more than 6 months.
Time Frame: Pre Treatment, 6 and 12 months Post Treatment
Population: The number analyzed in one or more rows differs from the overall number analyzed because not all patients had their EDSS evaluated and some patients were lost to followed up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation | Standard Therapy for MS
Number analyzed (Participants) | 52 | 54
units on a scale
  Pre Treatment | 3.4 (1.2) | 3.3 (1.0)
  6 Months Post Treatment | 2.5 (1.4) | 3.7 (1.5)
  12 Months Post Treatment: number analyzed (Participants) | 50 | 48
  12 Months Post Treatment | 2.4 (1.4) | 4 (1.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during transplant and at 1 year post Treatment
Arm/Group | Hematopoietic Stem Cell Transplantation | Standard Therapy for MS
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/55
Other Adverse Events (participants affected / at risk) | 17/52 | 0/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=52) | Standard Therapy for MS (N=55)
Febrile Neutropenia (culture negative) (General disorders) | 13 (13) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 17 (17) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 13 (13) | 0 (0)
Hypergylcemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations to the study are the relatively small number of patients who were treated compared with pharmaceutical sponsored trials, and the relatively small sample size resulted in small numbers of patients available to assess longer term outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes